CLINICAL TRIAL: NCT00890695
Title: Randomized Controlled Trial of an Outpatient Strategy of Ready to Use Supplementary Food (RUSF) Among Moderately Malnourished Children With Acute Infection
Brief Title: Effectiveness of Supplementary Feeding During Infection Among Moderately Malnourished Children
Acronym: MODMAL
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: New provision of supplementary feeds for moderately malnourished children
Sponsor: University of Oxford (Other)
Responsible Party: Principal Investigator, James Berkley, PI, University of Oxford
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SSC 1415
Record Dates: First submitted 2009-04-29; First posted 2009-04-30 (Estimated); Results first posted 2013-07-19 (Estimated); Last update posted 2017-08-14 (Actual); Status verified 2017-06

CONDITIONS: Malnutrition; Infection
Keywords: supplementary feeding; moderate malnutrition; acute infection; developing country; children
MeSH Terms: conditions — Malnutrition; Infections

STUDY DESIGN:
Intervention Model Description: Open label randomised trial of nutrition products
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ready to use supplementary food (RUSF) (Active Comparator): The RUSF intervention consists of a food paste made of maize, soya, sorghum, vegetable oil, sugar, dried skim milk and vitamin/mineral premix, prepared by VALID Nutrition in collaboration with Insta Products, Kenya in accordance with composition specified by the latest WHO expert consultation in 2008. Children in the intervention arm receive 4 weeks supply of RUSF. The amount supplied is based on the child's weight to give energy supplement of 100kcal per kg per day, equivalent to 25g RUSF per kg per day.
  Interventions: Dietary Supplement: Ready to use supplementary food (RUSF)
- Normal diet (standard of care) (No Intervention): For equity, parents or guardians of children in the usual diet arm will be given 2 bags of maize meal(4Kg) for family consumption instead of RUSF. All parents and carers in both arms will also receive standard nutritional advice as specified in the current WHO IMCI handbook.

INTERVENTIONS:
Dietary Supplement: Ready to use supplementary food (RUSF) — It is a strategy of detection of moderate malnutrition and providing advice and short term provision of a standard formulation of ready to use supplementary food (RUSF) for 4 weeks with appropriate counseling on its use.The amount supplied will be based on the child's weight; 100kcal per kg per day which is equivalent to 25g RUSF per kg per day.
  Other Names: RUSF
  Arms: Ready to use supplementary food (RUSF)

SUMMARY:
The purpose of this study is to determine whether an outpatient-based strategy of short-term, ready to use supplementary food (RUSF) among moderately malnourished children with acute infections achieves greater improvement in anthropometric measurements of wasting than usual diet.

DETAILED DESCRIPTION:
Under nutrition is a contributing factor to at least a third of child deaths. Whilst severe malnutrition has the highest mortality risk, most malnutrition-related deaths are thought to be related to mild-moderate malnutrition.This is because moderate malnutrition is common, it directly increases the risk of death from common infectious diseases and may progress to severe malnutrition.

Malnutrition may arise from poverty, food insecurity or inadequate nutrition being offered, and may begin early in life. Malnutrition is exacerbated by the multiple effects of infectious diseases such as gastroenteritis, pneumonia, malaria or HIV. All these common infections are associated with net protein loss with diversion of essential amino acids to producing acute phase and immune response proteins. Fever is associated with an increased resting energy expenditure of 7 to 13% per degree Centigrade. Activation of inflammatory cascades also causes reduced appetite and loss of lean tissue and fat. Acute infection is therefore associated with growth faltering, resulting in a vicious cycle. Acute infection is therefore a potential target for intervention to interrupt the vicious cycle between malnutrition and infection in children.

This study aims to evaluate a strategy of giving short-term RUSF as a supplement to usual diet at home, without daily observed feeding, administered through existing health services at Kilifi District Hospital, Kenya. RUSF has a very low moisture content and is essentially a lipid-enveloped paste, it is microbiologically stable with a long shelf life at tropical temperatures and preserves delicate micronutrients such as vitamin A.

ELIGIBILITY:
Inclusion Criteria:

* Age 6 months to 5 years
* Mid-upper arm circumference (MUAC) less than 12.5 cm
* Resident in the Kilifi demographic surveillance (DSS) area
* Presentation with acute (<5 days) illness including respiratory infection, malaria, diarrhoeal disease or other acute infection.
* If admitted, admission of <5 days, recruited at discharge.

Exclusion Criteria:

* Severe malnutrition (WHZ score < -3 or Kwashiorkor)
* Requiring admission to hospital in the opinion of clinician
* Known allergy to maize, soya, sorghum, milk or any RUSF components.
* Consent declined
* Underlying condition precluding assessment or inclusion
* Any other reason why the consenting investigator thinks it is not appropriate for them to take part.

Ages: 6 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 64 (Actual)
Dates: Start 2009-05; Primary Completion 2009-10 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James A Berkley, Principal Investigator — KEMRI-Wellcome Trust Collaborative Research Program
Locations (2):
- Kenya (2):
  - Kemri Wellcome Trust Research Programme, Kilifi, Coast Province
  - Kilifi District Hospital- OPD, Kilifi, Coast

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was started on June 5 2009 and finished on October 8 2009. The study was terminated early because of an inadequate recruitment rate and because a donor-funded supplementary feeding programme targeting moderately malnourished children was started in September 2009.
Pre-assignment Details: Of the 7,132 sick children aged 6 months to 5 years seen in outpatients during the study period, 190 with a mid upper arm circumference (MUAC) <12.5cm were assessed for eligibility. Randomization was carried out on 65 children who were eligible and whose carers consented. 1 was withdrawn: weight for height Z score (WHZ) was found to be <-3.
Groups:
- 1 Ready to Use Supplementary Food (RUSF): Products, Kenya. The RUSF composition is in accordance with recommended supplementary feed composition specified by the latest WHO expert consultation in 2008 reported by Golden et al. It is formulated to provide 507 kcal per 100g, 6% protein/energy ratio and 55% fat/energy ratio. Essential fatty acids contained are N-6 (linoleic acid) 6 kcal % and N-3 (o-linoleic) 0.3 kcal %. Vitamin and mineral premix (3%) will provide the currently recommended nutrient intake for moderately malnourished children of minerals (K, Na, Ca, P, Mg, Fe, Zn, Cu, Se, I, Mn, Cr, Mo, F), Vitamins (thiamine, riboflavin, pyridoxine, niacin, Vit B12, folic acid, Vit C, Biotin, Pantothenic acid, Vit A, Vit D,Vit E and Vit K).
  initial visit. The amount supplied is based on the child's weight; the recommended energy supplement being 100kcal per kg per day which is equivalent to 25g RUSF per kg per day.
- 2 Normal Diet: For equity, parents or guardians of children in the usual diet arm are given 2 bags of maize meal (4Kg) for family consumption instead of RUSF. All parents and carers in both arms will also receive standard nutritional advice as specified in the current WHO IMCI handbook.
Period: Overall Study
Arm/Group | 1 Ready to Use Supplementary Food (RUSF) | 2 Normal Diet
Started | 32 | 33
Completed | 31 | 33
Not Completed | 1 | 0
Not completed — Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- 1 RUSF: RUSF prescribed for the child for 4 weeks
- 2 Normal Diet: normal diet arm
- Total: Total of all reporting groups
Arm/Group | 1 RUSF | 2 Normal Diet | Total
Number analyzed (Participants) | 31 | 33 | 64
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 31 | 33 | 64
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 1.21 (0.55) | 1.15 (0.46) | 1.18 (0.50)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 23 | 49
  Male | 5 | 10 | 15
Region of Enrollment [Number; unit: participants]
  Kenya | 31 | 33 | 64

OUTCOME MEASURES:

1. Primary Outcome: Weight for Height z Score at 4 Weeks
Description: The primary endpoint is weight for height z scores (WHZ), calculated from weight and height measures with reference to the WHO growth standards 2006. WHZ is a measure of wasting and acute malnutrition.
  A WHZ of zero is the median value of the reference population. Negative scores indicate undernutrition. Moderate and severe acute malnutrition are defined as WHZ<-2 and <-3 respectively. These correspond to 2 and 3 standard deviations below the reference median.
  Of all the anthropometric measures in regular use, WHZ and mid upper arm circumference (MUAC) have the strongest associations with infectious disease incidence and risk of death. WHZ is more appropriate than Weight for Age (WAZ), which is normally used in growth monitoring, because WAZ measures a combination of wasting and stunting (chronic malnutrition). Stunting is unlikely to be affected by short term intervention. WHZ is assessed by anthropometry, following WHO guidelines.
Time Frame: between enrolment and 4 weeks
Population: All participants recruited until trial was halted
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | 1 RUSF | 2 Normal Diet
Number analyzed (Participants) | 31 | 33
units on a scale | -1.83 [-2.15 to -1.51] | -1.44 [-1.65 to -1.22]

2. Secondary Outcome: WHZ Score at 3 Months
Time Frame: between enrolment and 3 months
Population: All participants recruited until trial halted
Measure: Mean (95% Confidence Interval); unit: Z scores
Arm/Group | 1 RUSF | 2 Normal Diet
Number analyzed (Participants) | 31 | 33
Z scores | -1.43 [-1.68 to -1.18] | -1.29 [-1.56 to -1.03]

3. Secondary Outcome: MUAC for Age Z Score at 3 Months
Time Frame: between enrolment and 4 weeks and at 3 months
Population: All participants recruited until trial halted
Measure: Mean (95% Confidence Interval); unit: Z score
Arm/Group | 1 RUSF | 2 Normal Diet
Number analyzed (Participants) | 31 | 33
Z score | -1.71 [-1.99 to -1.43] | -1.62 [-1.95 to -1.28]

4. Secondary Outcome: Development of Severe Malnutrition (WHZ Score <-3 and/or Kwashiorkor)
Time Frame: at 4 weeks and 3 months
Population: All participants recruited until trial halted
Measure: Number; unit: participants
Arm/Group | 1 RUSF | 2 Normal Diet
Number analyzed (Participants) | 31 | 33
participants | 4 | 2

5. Secondary Outcome: Anemia (Hb <9.3g/dl)
Time Frame: at 4 weeks
Population: All participants recruited until trial halted
Measure: Number; unit: participants
Arm/Group | 1 RUSF | 2 Normal Diet
Number analyzed (Participants) | 31 | 33
participants | 16 | 11

6. Secondary Outcome: Hospital Admission or Death
Time Frame: from enrolment to 3 months
Population: All participants recruited until trial halted
Measure: Number; unit: participants
Arm/Group | 1 RUSF | 2 Normal Diet
Number analyzed (Participants) | 31 | 33
participants | 4 | 5

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | 1 RUSF | 2 Normal Diet
Serious Adverse Events (participants affected / at risk) | 4/31 | 5/32
Other Adverse Events (participants affected / at risk) | 0/31 | 0/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1 RUSF (N=31) | 2 Normal Diet (N=32)
Gastroenteritis (Gastrointestinal disorders) | 1 (2) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Severe malnutrition (Metabolism and nutrition disorders) | 2 (3) | 3 (3)

LIMITATIONS AND CAVEATS:
The trial was forced to stop early, 65 recruited. Analysis was inadequately powered to detect the changes in WHZ score and MUAC, the analysis of which had been originally planned for a sample size of 400.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes